CLINICAL TRIAL: NCT04975997
Title: A Phase 3, Two-Stage, Randomized, Multicenter, Open-label Study Comparing Iberdomide, Daratumumab and Dexamethasone (IberDd) Versus Daratumumab, Bortezomib, and Dexamethasone (DVd) in Subjects With Relapsed or Refractory Multiple Myeloma (RRMM)
Brief Title: Open-label Study Comparing Iberdomide, Daratumumab and Dexamethasone (IberDd) Versus Daratumumab, Bortezomib, and Dexamethasone (DVd) in Participants With Relapsed or Refractory Multiple Myeloma (RRMM)
Acronym: EXCALIBER-RRMM
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CC-220-MM-002; U1111-1260-2872 (Other: UTN Number); 2020-000431-49 (EudraCT Number)
Record Dates: First submitted 2021-07-02; First posted 2021-07-26 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-07

CONDITIONS: Multiple Myeloma
Keywords: Iberdomide; CC-220; Daratumumab; Darzalex Faspro; Bortezomib; Velcade; Dexamethasone; MM; Multiple Myeloma; RRMM; CELMoD; Cereblon Modulators
MeSH Terms: conditions — Multiple Myeloma | interventions — Dexamethasone; daratumumab; Bortezomib; iberdomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Daratumumab in combination with Iberdomide and dexamethasone - Dose 1 (Experimental): Participants will receive oral iberdomide, subcutaneous daratumumab and oral dexamethasone.
  Interventions: Drug: Dexamethasone; Drug: Daratumumab; Drug: Iberdomide
- Daratumumab in combination with Iberdomide and dexamethasone - Dose 2 (Experimental)
  Interventions: Drug: Dexamethasone; Drug: Daratumumab; Drug: Iberdomide
- Daratumumab in combination with Iberdomide and dexamethasone - Dose 3 (Experimental)
  Interventions: Drug: Dexamethasone; Drug: Daratumumab; Drug: Iberdomide
- Daratumumab in combination with dexamethasone and bortezomib (Active Comparator): Participants will receive subcutaneous daratumumab, bortezomib and oral dexamethasone
  Interventions: Drug: Dexamethasone; Drug: Bortezomib; Drug: Daratumumab

INTERVENTIONS:
Drug: Dexamethasone — Oral dexamethasone 40mg on days 1, 8, 15, 22 of a 28-day cycle
Drug: Daratumumab — Subcutaneous Daratumumab 1800mg on Days 1, 8, 15 and 22 for Cycles 1 to 2, on Days 1 and 15 for Cycles 3 to 6, and then on Day 1 for Cycle 7+ of a 28-day cycle
  Other Names: DARZALEX FASPRO
  Arms: Daratumumab in combination with Iberdomide and dexamethasone - Dose 1; Daratumumab in combination with Iberdomide and dexamethasone - Dose 2; Daratumumab in combination with Iberdomide and dexamethasone - Dose 3
Drug: Bortezomib — Subcutaneous Bortezomib 1.3 mg/m2 on Days 1, 4, 8 and 11 of each 21-day cycle for a total of 8 cycles.
  Arms: Daratumumab in combination with dexamethasone and bortezomib
Drug: Iberdomide — Oral Iberdomide 1.0mg on Days 1 to 21 of a 28-day cycle
  Other Names: CC-220; BMS-986382
  Arms: Daratumumab in combination with Iberdomide and dexamethasone - Dose 1
Drug: Iberdomide — Oral Iberdomide 1.3mg on Days 1 to 21 of a 28-day cycle
  Other Names: CC-220; BMS-986382
  Arms: Daratumumab in combination with Iberdomide and dexamethasone - Dose 2
Drug: Iberdomide — Oral Iberdomide 1.6mg on Days 1 to 21 of a 28-day cycle
  Other Names: CC-220; BMS-986382
  Arms: Daratumumab in combination with Iberdomide and dexamethasone - Dose 3
Drug: Dexamethasone — Oral dexamethasone 20mg on days 1,2, 4,5,8,9,11,12 of a 21-day cycle from cycles 1-8
  Arms: Daratumumab in combination with dexamethasone and bortezomib
Drug: Daratumumab — Subcutaneous daratumumab 1800mg Cycles 1 to 3 on Days 1, 8, 15 of a 21-day cycle, Cycles 4 to 8 on Day 1 of a 21-day cycle and Cycles 9+ on Day 1 of a 28-day cycle.
  Other Names: DARZALEX FASPRO
  Arms: Daratumumab in combination with dexamethasone and bortezomib

SUMMARY:
This is a multicenter, two-stage, randomized, controlled, open-label, Phase 3 study comparing the efficacy and safety of iberdomide in combination with dexamethasone and daratumumab (IberDd) versus daratumumab, bortezomib, and dexamethasone (DVd) in participants with relapsed or refractory multiple myeloma (RRMM).

DETAILED DESCRIPTION:
This is a multicenter, two-stage, randomized, controlled, open-label, Phase 3 study comparing the efficacy and safety of iberdomide in combination with dexamethasone and daratumumab (IberDd) versus daratumumab, bortezomib, and dexamethasone (DVd) in participants with relapsed or refractory multiple myeloma (RRMM). Approximately 200 patients randomized in stage 1 to one of three iberdomide dose levels of 1, 1.3, or 1.6 mg in combination with daratumumab and dexamethasone (Treatment Arms A1, A2, or A3), or to the DVd comparator arm (Treatment Arm B).

In Stage 2 of the study, approximately 664 additional subjects will be randomized 1:1 between 2 treatment arms:

* Approximately 332 subjects will be randomized to receive Treatment Arm A (IberDd)
* Approximately 332 subjects will be randomized to receive Treatment Arm B (DVd)

Participants in both treatment arms will continue to receive treatment until confirmed progressive disease (PD), unacceptable toxicity or withdrawal of consent. To ensure accuracy and completeness of the primary endpoint assessment of progression-free survival (PFS), participants who permanently discontinue study treatment for any reason, other than confirmed PD or withdrawal of consent, will continue to be followed for disease assessment.

The study will be conducted in compliance with International Council for Harmonisation (ICH) and Good Clinical Practices (GCPs).

ELIGIBILITY:
Inclusion Criteria

* Documented diagnosis of multiple myeloma (MM) and measurable disease.
* Received 1 to 2 prior lines of anti-myeloma therapy.
* Must have documented disease progression during or after their last anti-myeloma regimen.
* Eastern Cooperative Oncology Group (ECOG) performance status score of 0, 1 or 2.

Exclusion Criteria

* Any condition that confounds the ability to interpret data from the study.
* Has plasma cell leukemia, Waldenstrom's macroglobulinemia or POEMS syndrome (polyneuropathy, organomegaly, endocrinopathy, monoclonal protein, and skin changes), or clinically significant amyloidosis.
* Known central nervous system involvement with MM.
* Prior therapy with iberdomide.
* Other protocol-defined Inclusion/Exclusion criteria apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 864 (Estimated)
Dates: Start 2022-06-23 (Actual); Primary Completion 2026-03-18 (Estimated); Study Completion 2032-06-25 (Estimated)

PRIMARY OUTCOMES:
Progression-free Survival (PFS) | Up to approximately 5 years
  To compare the efficacy of iberdomide (also known as BMS-986382), daratumumab, and dexamethasone (IberDd) to that of daratumumab, bortezomib, and dexamethasone (DVd) in participants with relapsed or refractory multiple myeloma (RRMM) in terms of progression free survival (PFS).
Minimal Residual Disease (MRD) negative Complete Response (CR) at any time | Up to approximately 5 years
  To compare the efficacy of iberdomide (also known as BMS-986382), daratumumab, and dexamethasone (IberDd) to that of daratumumab, bortezomib, and dexamethasone (DVd) in participants with relapsed or refractory multiple myeloma (RRMM) in terms of minimal residual disease (MRD) negative complete response (CR) at any time.

SECONDARY OUTCOMES:
Overall Survival (OS) | Up to approximately 5 years
  To evaluate clinical efficacy in terms of overall survival (OS) in participants with relapsed or refractory multiple myeloma (RRMM) treated with iberdomide, daratumumab, and dexamethasone (IberDd) compared to daratumumab, bortezomib, and dexamethasone (DVd).
Sustainability of Minimal Residual Disease (MRD) negativity | Up to approximately 5 years
  To evaluate the sustainability of minimal residual disease (MRD) negativity.
Overall Response Rate (ORR) | Up to approximately 5 years
  Calculated as percentage of participants who achieve best response of partial response (PR) or better according to the IMWG Uniform Response Criteria for multiple myeloma.
Time to response (TTR) | Up to approximately 5 years
  Time from randomization to the first documentation of response (PR or better).
Duration of Response (DoR) | Up to approximately 5 years
  Time from the first documentation of response (PR or better) to the first documentation of progressive disease (PD) or death due to any cause, whichever occurs first.
Time to Progression (TTP) | Up to approximately 5 years
  The time from randomization to the first documented disease progression.
Time to Next Treatment (TTNT) | Up to approximately 5 years
  Time from randomization to the start of the next antimyeloma treatment.
Progression-free Survival 2 (PFS2) | Up to approximately 5 years
  Time from randomization to progression on the next anti-myeloma treatment or death due to any cause, whichever occurs first.
Safety | Up to approximately 5 years
  Type, frequency, seriousness and severity of adverse events (AEs), and relationship of AEs to study treatment.
European Organization for Research and Treatment of Cancer - Quality of Life C30 Questionnaire (EORTC QLQ-C30) | Up to approximately 5 years
  Mean changes from baseline in subscale scores in subject-reported health related quality of life outcomes and multiple myeloma-related symptoms as measured by the EORTC QLQ-C30.
European Quality of Life Multiple Myeloma Module (EORTC QLQ-MY20) | Up to approximately 5 years
  EORTC QLQ-MY20 is a 20-item myeloma module intended for use among participants varying in disease stage and treatment modality. Mean changes from baseline in subscale scores in subject-reported health related quality of life outcomes and multiple myeloma-related symptoms as measured by the EORTC QLQ- MY20.
Recommended iberdomide dose for Stage 2 | Up to approximately 1 year
Area under the plasma concentration-time curve from time zero to tau (AUC(TAU)) | Up to approximately 1 year
Maximum plasma concentration (Cmax) | Up to approximately 1 year
Time to maximum plasma concentration (Tmax) | Up to approximately 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (259):
- United States (43):
  - Local Institution - 035, Hot Springs, Arkansas
  - Local Institution - 641, Cerritos, California
  - Local Institution - 681, Fountain Valley, California
  - Local Institution - 047, Los Angeles, California
  - Local Institution - 684, Newport, California
  - Local Institution - 033, New Haven, Connecticut
  - Local Institution - 029, Fort Myers, Florida
  - Local Institution - 693, Ocala, Florida
  - Local Institution - 028, St. Petersburg, Florida
  - Local Institution - 045, Tamarac, Florida
  - Local Institution - 034, West Palm Beach, Florida
  - Local Institution - 685, Weston, Florida
  - Local Institution - 018, Atlanta, Georgia
  - Local Institution - 640, Elk Grove Village, Illinois
  - Local Institution - 697, Dyer, Indiana
  - Local Institution - 040, Louisville, Kentucky
  - Local Institution - 041, Alexandria, Louisiana
  - Local Institution - 682, Baton Rouge, Louisiana
  - Local Institution - 027, Baton Rouge, Louisiana
  - Local Institution - 698, Baltimore, Maryland
  - Local Institution - 014, Bethesda, Maryland
  - Local Institution - 688, Columbia, Maryland
  - Local Institution - 010, Boston, Massachusetts
  - Local Institution - 009, Worcester, Massachusetts
  - Local Institution - 645, Burnsville, Minnesota
  - Local Institution - 031, Kansas City, Missouri
  - Local Institution - 046, Billings, Montana
  - Local Institution - 015, Summit, New Jersey
  - Local Institution - 691, New York, New York
  - Local Institution - 039, Durham, North Carolina
  - Local Institution - 038, Cincinnati, Ohio
  - Local Institution - 037, Cleveland, Ohio
  - Local Institution - 008, Cleveland, Ohio
  - Local Institution - 036, Columbus, Ohio
  - Local Institution - 680, Tulsa, Oklahoma
  - Local Institution - 043, Portland, Oregon
  - Local Institution - 030, Chattanooga, Tennessee
  - Local Institution - 021, Nashville, Tennessee
  - Local Institution - 687, Austin, Texas
  - Local Institution - 695, Houston, Texas
  - Local Institution - 642, Newport News, Virginia
  - Local Institution - 643, Roanoke, Virginia
  - Local Institution - 025, Madison, Wisconsin
- Argentina (2):
  - Local Institution - 080, Ciudad Autanoma de Buenos Aires, Buenos Aires
  - Local Institution - 083, Villa Elisa, Buenos Aires
- Australia (12):
  - Local Institution - 813, Birtinya, Queensland
  - Local Institution - 812, Douglas, Queensland
  - Local Institution - 803, Adelaide, South Australia
  - Local Institution - 806, Bedford Park, South Australia
  - Local Institution - 802, Clayton, Victoria
  - Local Institution - 809, East Melbourne, Victoria
  - Local Institution - 801, Melbourne, Victoria
  - Local Institution - 811, Murdoch, Western Australia
  - Local Institution - 807, West Perth, Western Australia
  - Local Institution - 804, Camperdown
  - Local Institution - 800, Fitzroy
  - Local Institution - 808, Garran
- Austria (6):
  - Local Institution - 155, Graz
  - Local Institution - 154, Linz
  - Local Institution - 153, Salzburg
  - Local Institution - 156, Sankt Pölten
  - Local Institution - 150, Vienna
  - Local Institution - 151, Vienna
- Belgium (2):
  - Local Institution - 172, Bruges
  - Local Institution - 174, Brussels
- Brazil (9):
  - Local Institution - 056, Curitiba, Paraná
  - Local Institution - 050, Porto Alegre, Rio Grande do Sul
  - Local Institution - 058, Porto Alegre, Rio Grande do Sul
  - Local Institution - 051, Barretos, São Paulo
  - Local Institution - 054, Jaú, São Paulo
  - Local Institution - 055, São Paulo, São Paulo
  - Local Institution - 053, Rio de Janeiro
  - Local Institution - 057, São Paulo
  - Local Institution - 052, São Paulo
- Canada (9):
  - Local Institution - 111, Calgary, Alberta
  - Local Institution - 103, Edmonton, Alberta
  - Local Institution - 112, Surrey, British Columbia
  - Local Institution - 104, Saint John, New Brunswick
  - Local Institution - 110, St. John's, Newfoundland and Labrador
  - Local Institution - 101, Halifax, Nova Scotia
  - Local Institution - 109, Ottawa, Quebec
  - Local Institution - 108, Québec, Quebec
  - Local Institution - 107, Saskatoon, Saskatchewan
- China (25):
  - Local Institution - 141, Changsha, Hunan
  - Local Institution - 129, Nanchang, Jiangxi
  - Local Institution - 143, Xi'an, Shaanxi
  - Local Institution - 142, Shanghai, Shanghai Municipality
  - Local Institution - 145, Taiyuan, Shanxi
  - Local Institution - 144, Wenzhou, Zhejiang
  - Local Institution - 140, Beijing
  - Local Institution - 139, Beijing
  - Local Institution - 138, Beijing
  - Local Institution - 126, Changchun
  - Local Institution - 121, Chaoyang District
  - Local Institution - 135, Guangzhou
  - Local Institution - 136, Guangzhou
  - Local Institution - 128, Hangzhou
  - Local Institution - 120, Hangzhou, Zhejiang
  - Local Institution - 127, Harbin
  - Local Institution - 134, Nanjing
  - Local Institution - 132, Shanghai
  - Local Institution - 130, Shanghai
  - Local Institution - 131, Shenyang
  - Local Institution - 124, Suzhu
  - Local Institution - 133, Tianjin
  - Local Institution - 137, Wuhan
  - Local Institution - 125, Xi'an
  - Local Institution - 123, Zhengzhou
- Czechia (3):
  - Local Institution - 601, Brno
  - Local Institution - 600, Ostrava-Poruba
  - Local Institution - 602, Prague
- Denmark (3):
  - Local Institution - 371, Aalborg
  - Local Institution - 370, Odense
  - Local Institution - 372, Roskilde
- Finland (3):
  - Local Institution - 231, Turku, Southwest Finland
  - Local Institution - 230, Helsinki
  - Local Institution - 232, Oulu
- France (10):
  - Local Institution - 463, Argenteuil
  - Local Institution - 462, La Roche-sur-Yon
  - Local Institution - 451, Lille
  - Local Institution - 458, Nancy
  - Local Institution - 454, Nantes
  - Local Institution - 456, Paris
  - Local Institution - 452, Paris
  - Local Institution - 464, Pessac
  - Local Institution - 465, Rouen
  - Local Institution - 457, Toulouse
- Germany (6):
  - Local Institution - 308, Kiel, Schleswig-Holstein
  - Local Institution - 301, Frankfurt am Main
  - Local Institution - 300, Hamburg
  - Local Institution - 302, Hamburg
  - Local Institution - 305, Heidelberg
  - Local Institution - 304, Lübeck
- Greece (5):
  - Local Institution - 573, Pátrai, Achaea
  - Local Institution - 574, Pátrai, Achaia
  - Local Institution - 571, Athens
  - Local Institution - 572, Thessaloniki
  - Local Institution - 570, Thessaloniki
- India (6):
  - Local Institution - 932, Hyderabad, Andhra Pradesh
  - Local Institution - 930, Bangalore, Karnataka
  - Local Institution - 934, Ernākulam, Kerala
  - Local Institution - 933, Mumbai, Maharashtra
  - Local Institution - 935, Kolkata, West Bengal
  - Local Institution - 931, Puducherry
- Ireland (3):
  - Local Institution - 752, Cork
  - Local Institution - 750, Dublin
  - Local Institution - 751, Galway
- Israel (5):
  - Local Institution - 874, Afula, Northern District
  - Local Institution - 872, Haifa
  - Local Institution - 871, Jerusalem
  - Local Institution - 870, Tel Aviv
  - Local Institution - 873, Tel Litwinsky
- Italy (12):
  - Local Institution - 415, Rome, Lazio
  - Local Institution - 400, Bologna
  - Local Institution - 408, Catania
  - Local Institution - 414, Genova
  - Local Institution - 404, Milan
  - Local Institution - 410, Novara
  - Local Institution - 412, Pavia
  - Local Institution - 402, Pisa
  - Local Institution - 405, Reggio Calabria
  - Local Institution - 401, Roma
  - Local Institution - 403, San Giovanni Rotondo FG
  - Local Institution - 406, Udine
- Japan (21):
  - Local Institution - 900, Matsuyama, Ehime
  - Local Institution - 917, Higashi-Ibaraki-gun, Ibaraki
  - Local Institution - 919, Shimotsuga, Tochigi
  - Local Institution - 920, Nerima-ku, Tokyo
  - Local Institution - 918, Shinagawa-ku, Tokyo
  - Local Institution - 915, Chuo-shi, Yamanashi
  - Local Institution - 912, Aomori
  - Local Institution - 916, Chiba
  - Local Institution - 911, Fukuoka
  - Local Institution - 903, Kamogawa
  - Local Institution - 902, Kyoto
  - Local Institution - 910, Nagoya
  - Local Institution - 901, Nagoya
  - Local Institution - 905, Okayama
  - Local Institution - 907, Osaka
  - Local Institution - 908, Ōsaka-sayama
  - Local Institution - 913, Sapporo
  - Local Institution - 914, Sendai
  - Local Institution - 906, Shibuya-ku
  - Local Institution - 909, Shinagawa-ku, Tokyo
  - Local Institution - 904, Toyohashi
- Local Institution - 183, Guadalajara, Jalisco, Mexico
- Netherlands (3):
  - Local Institution - 351, Dordrecht, South Holland
  - Local Institution - 354, Amsterdam
  - Local Institution - 352, The Hague
- Norway (3):
  - Local Institution - 202, Bergen
  - Local Institution - 200, Oslo
  - Local Institution - 201, Trondheim
- Poland (6):
  - Local Institution - 631, Bialystok, Podlaskie Voivodeship
  - Local Institution - 633, Krakow
  - Local Institution - 635, Nowy Sącz
  - Local Institution - 634, Poznan
  - Local Institution - 630, Warsaw
  - Local Institution - 636, Wałbrzych
- Portugal (5):
  - Local Institution - 545, Coimbra
  - Local Institution - 543, Lisbon
  - Local Institution - 544, Lisbon
  - Local Institution - 540, Porto
  - Local Institution - 541, Porto
- South Korea (8):
  - Local Institution - 974, Daegu
  - Local Institution - 973, Gyeonggi-do
  - Local Institution - 975, Hwasun-gun
  - Local Institution - 971, Seoul
  - Local Institution - 976, Seoul
  - Local Institution - 972, Seoul
  - Local Institution - 970, Seoul
  - Local Institution - 977, Seoul
- Spain (17):
  - Local Institution - 514, Pamplona, Navarre
  - Local Institution - 505, Barcelona
  - Local Institution - 502, Barcelona
  - Local Institution - 511, Barcelona
  - Local Institution - 501, Cáceres
  - Local Institution - 509, Córdoba
  - Local Institution - 510, Madrid
  - Local Institution - 516, Madrid
  - Local Institution - 504, Madrid
  - Local Institution - 513, Madrid
  - Local Institution - 503, Málaga
  - Local Institution - 508, Murcia
  - Local Institution - 506, Oviedo
  - Local Institution - 515, Salamanca
  - Local Institution - 500, Santiago de Compostela
  - Local Institution - 512, Valencia
  - Local Institution - 507, Zaragoza
- Sweden (2):
  - Local Institution - 272, Borås
  - Local Institution - 271, Helsingborg
- Switzerland (2):
  - Local Institution - 851, Chur
  - Local Institution - 850, Sankt Gallen
- Taiwan (7):
  - Local Institution - 955, Niao-Sung Hsiang Kaohsiung County
  - Local Institution - 952, Taichung
  - Local Institution - 954, Taichung
  - Local Institution - 951, Tainan, Taiana
  - Local Institution - 950, Taipei
  - Local Institution - 956, Taipei, Zhongzheng Dist.
  - Local Institution - 953, Taoyuan
- Turkey (Türkiye) (9):
  - Local Institution - 778, Kavaklıdere, Ankara
  - Local Institution - 776, Yenimahalle, Ankara
  - Local Institution - 777, Pendik, Istanbul
  - Local Institution - 771, Balçova, İzmir
  - Local Institution - 775, Bornova, İzmir
  - Local Institution - 773, Samsun, Kurupelit
  - Local Institution - 770, Ankara
  - Local Institution - 772, Gaziantep
  - Local Institution - 774, Kayseri
- United Kingdom (11):
  - Local Institution - 702, Nottingham, Nottinghamshire
  - Local Institution - 705, Belfast Northern Ireland
  - Local Institution - 700, Birmingham
  - Local Institution - 707, Canterbury Kent
  - Local Institution - 704, Lancashire Blackpool
  - Local Institution - 701, London
  - Local Institution - 709, London
  - Local Institution - 706, Oxford
  - Local Institution - 711, Portsmouth
  - Local Institution - 713, Sutton
  - Local Institution - 708, Wolverhampton

IPD SHARING:
Plan to Share IPD: Yes
Information relating to our policy on data sharing and the process for requesting data can be found at the following link:
  https://www.celgene.com/research-development/clinical-trials/clinical-trials-data-sharing/
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: See Plan Description
Access Criteria: See Plan Description
URL: https://www.bms.com/researchers-and-partners/clinical-trials-and-research/disclosure-commitment.html

REFERENCES:
- [Derived] Lonial S, Dimopoulos MA, Berdeja JG, Richardson PG, Quach H, Rodriguez-Otero P, Maciag P, Hong K, Amatangelo M, Chen M, van de Donk NWCJ. EXCALIBER-RRMM: a phase III trial of iberdomide, daratumumab, and dexamethasone in relapsed/refractory multiple myeloma. Future Oncol. 2025 Jun;21(14):1761-1769. doi: 10.1080/14796694.2025.2501920. Epub 2025 May 10. PMID 40346992
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsclinicaltrials.com/us/en/clinical-trials/NCT04975997.html